CLINICAL TRIAL: NCT01917279
Title: A Randomized Phase III Study of Metronomic vs. Intermittent Capecitabine Maintenance Therapy Following First-line Capecitabine and Docetaxel Therapy in HER2-negative Metastatic Breast Cancer
Brief Title: Capecitabine Maintenance Therapy Following Capecitabine Combined With Docetaxel in Treatment of mBC
Acronym: CAMELLIA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Binghe Xu (Unknown)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Binghe Xu, Director of Medical Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28898
Record Dates: First submitted 2013-07-19; First posted 2013-08-06 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasms; Neoplasms by Site; Neoplasm Metastasis; Breast Diseases; Skin Diseases
Keywords: Metastatic Breast Cancer; Antineoplastic Agents; Therapeutic Uses; Antimetabolites; Tubulin Modulators; Maintenance chemotherapy; Metronomic chemotherapy; Capecitabine; Docetaxel
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Neoplasm Metastasis; Breast Diseases; Skin Diseases | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Capecitabine (Active Comparator): Capecitabine 1000 mg/m2 twice daily on days 1-14 of each 3-week cycle.
  Interventions: Drug: Docetaxel plus Capecitabine; Drug: Intermittent Capecitabine
- Metronomic Capecitabine (Experimental): Capecitabine 500 mg three times daily on days 1-21 of each 3-week cycle
  Interventions: Drug: Docetaxel plus Capecitabine; Drug: Metronomic Capecitabine

INTERVENTIONS:
Drug: Docetaxel plus Capecitabine — Eligible patients will receive treatment with Capecibatine (1000 mg/ m2 twice daily D1-14 Q3W) plus docetaxel(75 mg/m2, D1,Q3W) for a maximum of 6 cycles, or be treated until disease progression, unacceptable toxicity or patient request for withdrawal, whichever occurs first. Each cycle is 3 weeks in duration.
  For the the patients with SD, PR or CR after initiate treatment phrase will enter into maintenance treatment phase.
Drug: Intermittent Capecitabine — Capecitabine 1000 mg/m2 twice daily on days 1-14 of each 3-week cycle
  Other Names: Xeloda
  Arms: Intermittent Capecitabine
Drug: Metronomic Capecitabine — Capecitabine 500 mg three times daily on days 1-21 of each 3-week cycle
  Other Names: Xeloda
  Arms: Metronomic Capecitabine

SUMMARY:
It is a phase III trial to explore the efficacy and safety of metronomic chemotherapy with Capecitabine versus intermittent Capecitabine as maintenance therapy following first-line Capecitabine plus Docetaxel chemotherapy in treatment of HER2-negative metastatic breast cancer(mBC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures or treatment as confirmation of the patient's awareness and willingness to comply with the study requirements.
* Female patients aged ≥ 18 years.
* Histologically confirmed and documented HER2-negative metastatic breast cancer.
* Previously untreated first-line chemotherapy.
* Patients with at least one measurable lesion according to RECIST criteria at study entry.
* Documented ER/PgR status.
* Prior hormone therapy for metastatic disease is allowed but must stop before study entry.
* KPS>70.
* Life expectancy of ≥12 weeks

Exclusion Criteria:

* Previous chemotherapy for metastatic breast cancer.
* Prior adjuvant/neoadjuvant chemotherapy within 6 months prior to first study treatment administration.
* Prior (radical)radiotherapy for the treatment of metastatic disease or major surgical procedure within 28 days prior to the first study treatment,
* Inadequate bone marrow function: absolute neutrophil count (ANC): <1.5 x 109/L, platelet count<75 x 109/L or hemoglobin <100g/L.
* Inadequate liver or renal function, defined as:

  1. Serum (total) bilirubin >2 x the upper limit of normal (ULN) for the institution
  2. AST/SGOT or ALT/SGPT >2.5 x ULN (>5 x ULN in patients with liver metastases)
  3. ALP >2.5 x ULN at baseline (>5 x ULN in patients with liver metastases).
  4. Serum creatinine>140umol/L.
* Pregnant or lactating females.
* Her-2 positive (ICH +++ or FISH positive).
* Symptomatic cerebral parenchyma and/or leptomeningeal metastases.
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Pre-existing peripheral neuropathy ≥grade 1 according NCI CTCAE 4.0.
* Mental disease or other conditions affecting on the compliance of patients.
* Other serious disease or medical condition:

  1. History of uncontrolled seizures, CNS disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent.
  2. Congestive heart failure, or unstable angina, myocardial infarction within ≤6 months prior to the first study treatment, uncontrolled hypertension and high risk, uncontrolled arrhythmias.
  3. Uncontrolled acute infection
* Inability to take or absorption oral medications.
* Concurrent or within 30 days using drugs of other clinical trials.
* Previous treatments containing Capecitabine (whether adjuvant or palliative treatment).
* Previous treatments containing docetaxel within 12 months.
* Known hypersensitivity to any of the study treatments or excipients.
* Any other conditions the research consider not appropriate to take part in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2013-10; Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 36 months
  Time from randomization to progression or death (whichever occurred first).

SECONDARY OUTCOMES:
Adverse events (AEs) | up to 36 months
  Adverse events (AEs) and laboratory tests graded according to the NCI CTCAE (version 4.0), premature withdrawals and vital signs. Hand-foot syndrome and diarrhea will be specially interested.
  Adverse events of special interest: hand-foot syndrome and diarrhea. The estimated HFS rate will be about 60% from intermittent Capecitabine vs about 10% from metronomic Capecitabine, diarrhea rate will be about 50% from intermittent Capecitabine vs about 10% from metronomic Capecitabine.
Overall survival (OS): | up to 52 months
  Time from randomization to death
Overall Response rates (ORR) | up to 36 months
  Defined as CR+PR, assessed based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria. It will be evaluated in the initial treatment phase and the maintenance treatment phase.
Clinical Benefit rate (CBR) | up to 36 months
  Defined as CR+PR+SD, assessed based on on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria. It will be evaluated in the initial treatment phase and the maintenance treatment phase
Time to Progression (TTP) | up to 36 months
  Time from randomization to disease progression
QoL | up to 36 months
  Using the EORTC quality of life questionnaire QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy Of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Yi Z, Feng K, Lv D, Guan Y, Shao Y, Ma F, Xu B. Genomic landscape of circulating tumor DNA in HER2-low metastatic breast cancer. Signal Transduct Target Ther. 2024 Dec 9;9(1):345. doi: 10.1038/s41392-024-02047-0. PMID 39648226
- [Derived] Guan X, Ma F, Li C, Wu S, Hu S, Huang J, Sun X, Wang J, Luo Y, Cai R, Fan Y, Li Q, Chen S, Zhang P, Li Q, Xu B. The prognostic and therapeutic implications of circulating tumor cell phenotype detection based on epithelial-mesenchymal transition markers in the first-line chemotherapy of HER2-negative metastatic breast cancer. Cancer Commun (Lond). 2019 Jan 3;39(1):1. doi: 10.1186/s40880-018-0346-4. PMID 30606259